CLINICAL TRIAL: NCT04653883
Title: Prognostic Impact of Sleep Disorders in Patients With Heart
Brief Title: Prognostic Impact of Sleep Disorders in Patients : Pro-TSIC Study
Acronym: Pro-TSIC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0307
Record Dates: First submitted 2020-09-04; First posted 2020-12-04 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure; Sleep Disorder; Insomnia
MeSH Terms: conditions — Heart Failure; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heart failure (HF) is a common and progressive condition associated with significant morbidity and mortality. Only 25-35% of patients survive 5 years after diagnosis.Sleep disorders are frequently found in this population with up to 94% of patients complaining of sleep disorders. Of these, insomnia and sleep disorders are the most common. The frequency of restless legs syndrome (RLS) varies between 4 and 40% depending on the studies. Patients with HF frequently experience poor sleep quality which is associated with deterioration in quality of life, alertness, and mood.

Few studies have examined the prognostic impact of sleep disturbances in this population. A greater morbidity and mortality is observed in the event of poor quality sleep or in the presence of sleep breathing disorders .

The investigators therefore propose to evaluate the sleep disorders of patients with HF by self-administered questionnaires, hypothesizing that complaints of poor sleep are linked to a poorer cardiovascular prognosis.

ELIGIBILITY:
Inclusion criteria:

- heart failure according to the 2016 criteria of the European Society of Cardiology.

Exclusion criteria:

- age less than 30 years

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in this study are the patients followed in the Cardiology Department of the Montpellier University Hospital and diagnosed with heart failure according to the 2016 criteria of the European Society of Cardiology.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
To study the occurrence of cardiovascular events, whether fatal or not, according to the presence or absence of sleep or wakefulness disorders | 1 day
  composite endpoint including mortality from any cause, hospitalization forrom any cardiovascular eventscause, heart transplantation and implantation of a defibrillator or circulatory assistance

SECONDARY OUTCOMES:
Evaluate the occurrence of fatal events according to the presence or absence of sleep or wakefulness disorders | 1 day
  Evaluate the occurrence of fatal events according to the presence or absence of sleep or wakefulness disorders
Evaluate the occurrence of cardiovascular non-fatal major adverse cardiovascular events according to the presence or absence of sleep or wakefulness disorders | 1 day
  Evaluate the occurrence of cardiovascular non-fatal major adverse cardiovascular events according to the presence or absence of sleep or wakefulness disorders
Evaluate the occurrence of fatal or non-fatal major adverse cardiovascular events depending on whether or not medication is taken for sleep disorders | 1 day
  Evaluate the occurrence of fatal or non-fatal major adverse cardiovascular events depending on whether or not medication is taken for sleep disorders

CONTACTS AND LOCATIONS:
Overall Officials: François BUGHIN, PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC